CLINICAL TRIAL: NCT01307371
Title: Effects and Mechanism of Autologous Bone Marrow Mononuclear Cells (BMMNC)Transplantation in Diabetic Patients With ST-Segment Elevation Myocardial Infarction (STEMI) Who Have Undergone Percutaneous Coronary Intervention (PCI)
Brief Title: Cell Therapy in Diabetic Patients With ST-Segment Elevation Myocardial Infarction(STEMI)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Department of Cardiovascular medicine, Xijing Hospital, Fourth Military Medical University
Other Study IDs: DIABETES-STEMI
Record Dates: First submitted 2011-02-24; First posted 2011-03-02 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2011-02

CONDITIONS: Left Ventricular Function Systolic Dysfunction; Left Ventricular Function Diastolic Dysfunction; Death; Myocardial Reperfusion Injury
Keywords: Bone Marrow Mononuclear cells;; Diabetes;; ST-segment Elevation Myocardial Infarction;; Percutaneous Coronary Intervention;; Left Ventricular Function
MeSH Terms: conditions — Death; Myocardial Reperfusion Injury; Diabetes Mellitus; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Diabetes: Patients with diabetes.
- non-diabetes: Patients without diabetes.

SUMMARY:
The purpose of this study is to investigate the efficacy and mechanism of bone marrow mononuclear cells (BMMNC) transplantation for diabetic and non-diabetic patients with ST-segment elevation myocardial infarction (STEMI)who have undergone percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
Stem cells are capable of the important properties of self-renewal and differentiation plasticity. Human autologous bone marrow mononuclear cells (BMMNC) contain CD34+ haematopoietic and CD34- mesenchymal stem cells. Both of these cell types may contribute to heart muscle repair in acute myocardial infarction (AMI). In recent years, a variety of clinical trials have explored the hypothesis that BMMNC transplantation may enhance the recovery of left ventricular function after AMI. The use of BMMNC is clinically justified and ethically unquestionable because no severe side effects have been reported and immunosuppressive therapy is unnecessary. More over, our previous work showed that patients without diabetes may benefit more from BMMNC transplantation. Thus, the aim of the present study was to investigate the efficacy and mechanism of bone marrow mononuclear cells (BMMNC) transplantation for diabetic and non-diabetic patients with ST-segment elevation myocardial infarction (STEMI)who have undergone PCI.

ELIGIBILITY:
Inclusion Criteria:

* age between 25 and 60 years old
* STEMI according to the WHO definition
* PCI <12 hours from the onset of symptoms
* LAD disease with an open infarct related artery

Exclusion Criteria:

* previous myocardial infarction (MI)
* cardiomyopathy
* atrial fibrillation or flutter
* previous heart surgery
* severe valvular heart disease
* disease of the hematopoietic system
* NYHA functional class IV heart failure at baseline
* severe renal, lung and liver disease
* cancer
* intra-cardiac thrombus
* bone marrow disease

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients of STEMI with the culprit lesion of left anterior decending (LAD)coronary artery were enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Number of patient death during the follow up period | 4years
  Number of patient death during the follow up period as a measure of safety

SECONDARY OUTCOMES:
Left ventricular ejection fraction | 4 years
  Left ventricular ejection fraction as evaluated by echocardiography and SPECT
Myocardial perfusion scores as evaluated by Single-photon emission computed tomography (SPECT) | 4 years
Infarct size as evaluated by Single-photon emission computed tomography (SPECT) | 4 years
Number of target vessel revascularization | 4 years
  Number of target vessel revascularization during the follow up period
Angina class according to the canadian cardiovascular society (CCS) classification | 4 years
Scores on the Seattle angina questionnaire | 4 years
six-min walk distance (6MWD) | 4 years
  Quality of life as evaluated by 6-min walk distance

CONTACTS AND LOCATIONS:
Overall Officials: Feng Cao, MD, PhD, Principal Investigator — Air Force Military Medical University, China
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China